

## Study Flow Diagram

Official Title: Double-Blind, Placebo-Controlled, Parallel-Group Randomized Controlled Trial to Evaluate the Efficacy and Safety of Nimsai Herbal in Patients with Grade 2-3 Hemorrhoids

NCT Number: NCT07034820

Protocol Number: NA-2024-001

Document Date: November 15, 2021

Sponsor: Nimsai Academia Bursa, Türkiye

Principal Investigator: Cem Atabiner Nimsai Academia

Phone: +90 532 459 3292

Email: cem.atabiner@kecioutdoor.com.tr

Prepared by: Nimsai Academia Bursa, Türkiye

Submission Format: PDF/A

Confidentiality Statement: This document contains confidential information and is intended solely for authorized personnel, investigators, and regulatory authorities. Unauthorized reproduction or distribution is prohibited. No participant names or identifiable information are included.

Citation: Hopewell S, Chan AW, Collins GS, Hróbjartsson A, Moher D, Schulz KF, et al. CONSORT 2025 Statement: updated guideline for reporting randomised trials. BMJ. 2025; 388:e081123. https://dx.doi.org/10.1136/bmj-2024-081123

© 2025 Hopewell et al. This is an Open Access article distributed under the terms of the Creative Commons Attribution License (<a href="https://creativecommons.org/licenses/by/4.0/">https://creativecommons.org/licenses/by/4.0/</a>), which permits unrestricted use, distribution, and reproduction in any medium, provided the original work is properly cited.



## **CONSORT 2025 Flow Diagram**

Flow diagram of the progress through the phases of a randomised trial of two groups (that is, enrolment, intervention allocation, follow-up, and data analysis)



Citation: Hopewell S, Chan AW, Collins GS, Hróbjartsson A, Moher D, Schulz KF, et al. CONSORT 2025 Statement: updated guideline for reporting randomised trials. BMJ. 2025; 388:e081123. https://dx.doi.org/10.1136/bmj-2024-081123

© 2025 Hopewell et al. This is an Open Access article distributed under the terms of the Creative Commons Attribution License (<a href="https://creativecommons.org/licenses/by/4.0/">https://creativecommons.org/licenses/by/4.0/</a>), which permits unrestricted use, distribution, and reproduction in any medium, provided the original work is properly cited.